CLINICAL TRIAL: NCT01853553
Title: Mineralocorticoid Antagonism and Endothelial Dysfunction in Autosomal Dominant Polycystic Kidney
Brief Title: Mineralocorticoid Antagonism and Endothelial Dysfunction in Autosomal Dominant Polycystic Kidney Disease (ADPKD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 13-1440; R01DK097081 (NIH)
Record Dates: First submitted 2013-05-08; First posted 2013-05-15 (Estimated); Results first posted 2019-08-20 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: ADPKD
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant | interventions — Spironolactone; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (2):
- Spironolactone (Experimental): Active arm
  Interventions: Drug: Spironolactone
- Sugar Pill (Placebo Comparator): Placebo
  Interventions: Drug: Sugar pill

INTERVENTIONS:
Drug: Spironolactone — Blood pressure medication.
  Arms: Spironolactone
Drug: Sugar pill — Placebo.
  Arms: Sugar Pill

SUMMARY:
The proposed research will determine the effectiveness of blocking aldosterone for improving the health and function of arteries in patients with autosomal dominant polycystic kidney disease (ADPKD). The study also will provide insight into how blocking aldosterone improves artery health by determining the physiological mechanisms (biological reasons) involved. Overall, the proposed research will provide important new scientific evidence upon which physicians can base recommendations to patients with ADPKD to decrease risk of developing cardiovascular diseases.

DETAILED DESCRIPTION:
Background: Cardiovascular complications are currently the major causes of mortality among patients with autosomal dominant polycystic kidney disease (ADPKD). Therefore, testing valid interventions to reduce morbidity and mortality within this population is of high priority. It is well documented that endothelial dysfunction coupled with abnormalities in markers of oxidative stress and inflammation develops early in ADPKD even before there is a significant decline in kidney function. Aldosterone levels are increased in patients with ADPKD and may contribute to cardiovascular disease by impairing endothelial function, and reducing vascular compliance. Of note, aldosterone antagonists have been shown to improve endothelial dysfunction in a number of studies in other patient populations. However, there has been no clinical interventional studies specifically targeting endothelial dysfunction in ADPKD. Our main goal is to establish the efficacy of an aldosterone antagonist (spironolactone) for treating vascular endothelial dysfunction and large elastic artery stiffness in ADPKD patients with preserve kidney function. A key secondary goal is to determine the integrative physiological (i.e., whole limb/artery to molecular) mechanisms underlying the beneficial effects of spironolactone.

Working Hypotheses:

1. Six months of an aldosterone antagonist will increase endothelium-dependent dilation (EDD) and reduce large elastic artery stiffness in ADPKD patients with preserve kidney function.
2. The improvements in EDD after aldosterone antagonist will be associated with reduced circulating and endothelial cell markers of oxidative stress and inflammation.
3. The improvements in large elastic artery stiffness after aldosterone antagonist will be associated with reduced circulating and endothelial cell markers of oxidative stress and inflammation, and changes in markers of structural protein turnover.

Impact on the Field: The expected results will provide the first insight into the:

* Efficacy of an aldosterone antagonist for the primary treatment of vascular dysfunction in ADPKD patients with preserve kidney function.
* Cellular and molecular physiological mechanisms by which these treatment benefits are conferred.

ELIGIBILITY:
Inclusion Criteria:

* Aged 20-55 years;
* Adults with ADPKD diagnosis based on Ravine criteria aged ≥ 30 years
* Estimated glomerular filtration rate ≥ 60 ml/min/1.73m2
* Hypertension defined as a systolic BP > 130 mm Hg and/or diastolic BP > 80 mmHg based on 3 separate measurements within the past year and currently on a minimum dose of an angiotensin converting enzyme inhibitor (minimum dose 10 mg P.O qd) or angiotensin receptor blocker (i.e., Losartan 25 mg P.O qd)
* If using antioxidants and/or omega-3 fatty acids, must discontinue 4 weeks prior to participation
* Free from alcohol dependence or abuse
* Mini-mental state examination score ≥ 24; ability to provide informed consent
* BMI < 40 kg/m2 (FMD measurements can be inaccurate in severely obese patients)
* Not taking medications that interact with agents administered during experimental sessions (e.g., sildenafil interacts with nitroglycerin)

Exclusion Criteria:

* • Average serum potassium >5.5 millequivalents or any single serum potassium > 6.0 millequivalents within the previous 6 months

  * Receiving an aldosterone antagonist within the previous 6 months
  * Use of a potassium sparing diuretic or any other drug that could contribute to hyperkalemia
  * Uncontrolled hypertension
  * Current smokers or history of smoking in the past 12 months
  * History of liver disease
  * History of heart failure (EF < 35%)
  * History of hospitalizations within the last 3 months
  * Active infection or antibiotic therapy
  * Warfarin use
  * Immunosuppressive therapy within the last year
  * Pregnancy

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2013-07; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michel B Chonchol, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- UColorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nowak KL, Gitomer B, Farmer-Bailey H, Wang W, Malaczewski M, Klawitter J, You Z, George D, Patel N, Jovanovich A, Chonchol M. Mineralocorticoid Antagonism and Vascular Function in Early Autosomal Dominant Polycystic Kidney Disease: A Randomized Controlled Trial. Am J Kidney Dis. 2019 Aug;74(2):213-223. doi: 10.1053/j.ajkd.2018.12.037. Epub 2019 Feb 23. PMID 30803706

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants were enrolled at the University of Colorado Denver Anschutz Medical Campus between July 2014 and June 2016 (the trial concluded according to enrollment determined by power calculations described below).Although Grant was awarded in 2013, recruitment did not start until 2014.
Pre-assignment Details: Participants were excluded if they had an average serum potassium >5.5 mEq/l or any single value >6.0 mEq/l in the past 6 months, received an aldosterone antagonist in the past 6 months, and were using a potassium sparing diuretic or other medication that could contribute to hyperkalemia.
Groups:
- Spironolactone: Active arm
  Spironolactone
  Participants were then randomized by the study coordinator according to a computer-generated random allocation sequence and received either the mineralocorticoid antagonist spironolactone or matching placebo. Participants were dosed at 25 mg/day for 4 weeks, with dosing escalated to 50 mg/day for the remainder of the study if tolerated by an individual participant.
- Sugar Pill: Placebo
  Sugar pill
Period: Overall Study
Arm/Group | Spironolactone | Sugar Pill
Started | 29 | 32
Completed | 28 | 32
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Spironolactone | Sugar Pill | Total
Number analyzed (Participants) | 29 | 32 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (10) | 34 (9) | 34 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 20 | 33
  Male | 16 | 12 | 28

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Flow Mediated Dilation at 6 Months.
Description: FMD will be determined using high-resolution ultrasonography
Time Frame: Baseline and 6 months.
Measure: Mean (Standard Deviation); unit: Percent change.
Groups:
- Spironolactone: Active arm
  Spironolactone
Arm/Group | Spironolactone | Sugar Pill
Number analyzed (Participants) | 28 | 32
Percent change. | -0.2 (3.2) | -0.4 (4.7)

2. Secondary Outcome: Change From Baseline in Vascular Stiffness at 6 Months.
Description: Aortic pulse wave velocity, a measure of large elastic arterial stiffness, and carotid compliance, a measure of large artery distensibility, will be determined. A transcutaneous custom tonometers (Noninvasive Hemodynamics Workstation, Cardiovascular Engineering Inc., Norwood, MA) will be positioned at the aorta and femoral artery to measure pulse wave velocity, and carotid artery compliance (and the β-stiffness index, a more blood pressure independent measure of local arterial stiffness) will be measured non-invasively using simultaneous high-resolution ultrasonography and applanation tonometry). Higher values correspond to greater stiffness.
Time Frame: Baseline and 6 months
Measure: Median (Standard Deviation); unit: m/s
Arm/Group | Spironolactone | Sugar Pill
Number analyzed (Participants) | 28 | 32
m/s | -37 (78) | -1 (89)

3. Other Pre Specified Outcome: Change in Circulating Markers of Oxidative Stress at 6 Months.
Description: All markers of oxidative stress will be assayed by multiplexed validated liquid chromatography (LC)/ LC-mass spectrometry (MS)/ MS.
Time Frame: Baseline and 6 months.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Spironolactone: Active arm
  Spironolactone 25 mg once daily.
- Sugar Pill: Placebo
  Sugar pill-1 tablet once daily.
Arm/Group | Spironolactone | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/32
Other Adverse Events (participants affected / at risk) | 0/28 | 0/32

LIMITATIONS AND CAVEATS:
A potential limitation to the study is a relatively small sample size; however, we were appropriately powered to detect an improvement in the primary endpoint given expected vascular endothelial function at the time the trial was designed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes